CLINICAL TRIAL: NCT03345381
Title: Impact of Breathing Exercises and Meditation on Health-Related Quality of Life in Dry Eye Disease Patients: A Pilot Study
Brief Title: Impact of Breathing Exercises and Meditation on Quality of Life in Dry Eye Disease Patients: A Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 110762
Record Dates: First submitted 2017-11-14; First posted 2017-11-17 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Depression; Quality of Life; Dry Eye; Anxiety; Sleep
MeSH Terms: conditions — Depression; Dry Eye Syndromes; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SKY + ASTM + usual care (Experimental): Sudarshan Kriya Yoga (SKY) followed by Automatic Self Transcending Meditation (ASTM) plus usual care
  Interventions: Other: SKY + ASTM + usual care
- Usual Care (Active Comparator): Treatment as usual
  Interventions: Other: Usual care

INTERVENTIONS:
Other: SKY + ASTM + usual care — Sudarshan Kriya Yoga (SKY) followed by Automatic Self Transcending Meditation (ASTM) involves breathing exercise followed by meditation.
  Arms: SKY + ASTM + usual care
Other: Usual care — Treatment as usual
  Arms: Usual Care

SUMMARY:
People staring at computer screens for long hours, blinking less frequently, or having long-term contact lens wear are prone to dry eye disease (DED). DED is a multifactorial disease accompanied by inflammation of the ocular surface. Further, DED may degrade vision and is associated with depression and have an adverse impact on patient's quality of life. Sudarshan Kriya Yoga (SKY) incorporates standardized collection of breathing techniques followed by Automatic Self Transcending Meditation (ASTM) may help reduce stress, depression, and anxiety, enhance quality of life in patients diagnosed with DED. Thus, the investigators will be studying the effect of SKY plus ASTM on quality of life of DED patients. The investigators plan to conduct a single-center pilot RCT. Patients with DED will be randomized to SKY followed by ASTM plus Usual care (UC) or UC alone to assess changes in health-related quality of life (HRQOL). HRQOL is a vital construct focusing on impact of health on quality of life. Along with HRQOL the investigators will measure changes in extent of depression and anxiety. Additionally, majority of current ophthalmic literature describes changes in clinical variables whilst lacking information on HRQOL. Thus, there is a high necessity to assess if there is an association between HRQOL and routinely measured clinical data. Through this study the investigators shall attempt to correlate HRQOL with clinical data.

DETAILED DESCRIPTION:
Background: Prevalence of dry eye disease (DED) ranges from 3.5% to 33.7% and increase with age. Further, DED is associated with decreased productivity, absenteeism from work, depression, and has an adverse impact on patient's quality of life. Odds of a DED patient suffering from depression is 2.9 and anxiety is 2.8. Yoga - a practice to help improve health and well-being - has also been the subject of clinical studies globally. Two central aspects of yoga practice are physical postures and breathing exercises. These breathing exercises aim to focus the mind, facilitate relaxation and enhance wellness.

Evidence further suggests beneficial effects of a standardized collection of breathing techniques called Sudarshan Kriya Yoga (SKY) on individuals suffering from depression. SKY includes three-stage breathing with Victory breath (slow deep breathing that consists of 4 to 6 breaths per minute), Bellow's breath (forceful rapid deep breathing that consists of 20 to 30 breaths per minute), and a rhythmic breath technique. SKY followed by Automatic Self Transcending Meditation (ASTM) involves breathing exercise followed by meditation. ASTM utilizes a specific sound value mantra to draw attention inward and permit the mind to experience a restful but alert state of consciousness. It helps quiet the mind and induces physiological and mental relaxation whilst the eyes are shut. ASTM may help with depression, anxiety, stress, and may enhance quality of life. Thus, the investigators will be studying the effect of SKY plus ASTM on quality of life of DED patients. Key goal of proposed research is to evaluate HRQOL, depression, anxiety of patients with DED in SKY followed by ASTM and usual care (UC) versus UC alone from baseline to 24 weeks.

Primary Hypothesis: The investigators hypothesize that in patients with dry eye disease in SKY + ASTM + UC may lead to significant improvement in HRQoL compared to UC alone from baseline to 24 weeks.

Secondary Hypotheses: The investigators hypothesize that in patients with DED 1) HRQoL is associated with regularly measured clinical variables 2) SKY + ASTM + UC leads to significant improvement in depression and anxiety symptoms at 24 weeks compared to UC alone.

ELIGIBILITY:
Inclusion Criteria:

* dry eye disease suspects or have mild to severe dry eye disease
* at least between 18 to 80 years of age
* deemed competent such as no language issues or communication barriers, no self-reported or physician diagnosed mental health disorder besides having depressive and anxiety symptoms
* have sufficient hearing to be able to follow verbal instructions and able to sit without physical discomfort for 30 minutes
* willing and able to attend 3 initial SKY and 4 initial ASTM training sessions
* willing to dedicate 20 minutes per day for SKY and 20 minutes twice per day to ASTM practice at their own home.

Exclusion Criteria:

* actively suicidal as per self-report (or score on CES-D) or on assessment by the physician
* they are currently participating in other similar studies
* currently practicing any type of formal meditation techniques regularly
* unable or unwilling to answer survey questions.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-07-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life (HRQoL) | Up to 24 weeks
  Health Related Quality of LIfe (HRQoL) is an essential measure of quality of life related to health. HRQoL will be measured using time trade-off (TTO) questionnaire. HRQoL varies between 0 and 1 where the score of 1 represents perfect health and 0 represents death.

SECONDARY OUTCOMES:
Visual Function Score | Up to 24 weeks
  Visual related quality of life measured using National Eye Institute Visual Function Questionnaire-25 (NEI VFQ-25). The most widely used instrument in vision-related functioning is the NEI VFQ-25. It was designed specifically for a clinical setting and consists of 12 domains: general health, general vision, visual pain, near activities, distance activities, social functioning, mental health, role difficulties, dependency, driving, colour vision and peripheral vision. The shorter 25-item version questionnaire is widely used in different groups of patients and shown to be internally consistent, reproducible and responsive in glaucoma patients. The NEI VFQ-25 scores have a closer relationship to clinical outcomes, in comparison to generic instruments. The scores range from 0 to 100 where higher score represents better vision related quality of life.
Depression | Up to 24 weeks
  Center for Epidemiologic Studies Depression Scale (CES-D) will be used to measure depression. It is one of the most common validated tools used to measure depression in research to identify depressive symptoms. Additionally, it is a brief standardized valid tool for assessing depressive symptoms. Possible range of scores is zero to 60, with the higher scores indicating the presence of more depressive symptoms.
State and Trait Anxiety | Up to 24 weeks
  State-Trait Anxiety Inventory (STAI)
Sleep Quality | Up to 24 weeks
  Pittsburgh Sleep Quality Index (PSQI)
Community Integration | Up to 24 weeks
  The community integration questionnaire (CIQ) was used to provide a quantitative indicator for the level of social support and ability to perform appropriate roles at home and within the community. The CIQ contains 15-items and uses behavioural items of integration to achieve better reliability. The total CIQ score ranges from 0 to 29, with a higher score representing a higher level of social support and complete community integration.
Canadian Dry Eye Assessment | Up to 24 weeks
  Canadian Dry Eye Assessment
Dry Eye Assessment | Up to 24 weeks
  Standardized Patient Evaluation of Eye Dryness (SPEED) Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Monali Malvankar, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- St. Joseph's Hospital, Ivey Eye Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
De-identified IPD collected in this study will not be available to other researchers (e.g. outside the primary research group). Because the primary research group has the necessary expertise to conduct analysis and do not need any outside help.

REFERENCES:
- [Background] Schein OD, Munoz B, Tielsch JM, Bandeen-Roche K, West S. Prevalence of dry eye among the elderly. Am J Ophthalmol. 1997 Dec;124(6):723-8. doi: 10.1016/s0002-9394(14)71688-5. PMID 9402817
- [Background] Schaumberg DA, Dana R, Buring JE, Sullivan DA. Prevalence of dry eye disease among US men: estimates from the Physicians' Health Studies. Arch Ophthalmol. 2009 Jun;127(6):763-8. doi: 10.1001/archophthalmol.2009.103. PMID 19506195
- [Background] Schaumberg DA, Sullivan DA, Buring JE, Dana MR. Prevalence of dry eye syndrome among US women. Am J Ophthalmol. 2003 Aug;136(2):318-26. doi: 10.1016/s0002-9394(03)00218-6. PMID 12888056
- [Background] Yu J, Asche CV, Fairchild CJ. The economic burden of dry eye disease in the United States: a decision tree analysis. Cornea. 2011 Apr;30(4):379-87. doi: 10.1097/ICO.0b013e3181f7f363. PMID 21045640
- [Background] Wan KH, Chen LJ, Young AL. Depression and anxiety in dry eye disease: a systematic review and meta-analysis. Eye (Lond). 2016 Dec;30(12):1558-1567. doi: 10.1038/eye.2016.186. Epub 2016 Aug 12. PMID 27518547
- [Background] Elder C, Nidich S, Moriarty F, Nidich R. Effect of transcendental meditation on employee stress, depression, and burnout: a randomized controlled study. Perm J. 2014 Winter;18(1):19-23. doi: 10.7812/TPP/13-102. PMID 24626068
- [Background] Burns JL, Lee RM, Brown LJ. The effect of meditation on self-reported measures of stress, anxiety, depression, and perfectionism in a college population. Journal of College Psychotherapy 25(2): 132-144, 2011.